CLINICAL TRIAL: NCT06742762
Title: A Phase I, Multicentre, Single-Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD5004
Brief Title: A Phase I Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD5004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7260C00006
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Renal Impairment
Keywords: Renal Impairment; Healthy participants; AZD5004; Pharmacokinetics; Safety
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Up to three groups (two renal impairment groups and controls with normal renal function) will be enrolled into this study.
  All subjects will receive the study intervention:
  Group 1 will enroll 7 participants with severe renal impairment Group 2 will enroll ~7 participants with normal renal function matched by sex, age, and body weight Group 3 (optional) will enroll 7 participants with moderate renal impairment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants with severe renal impairment will receive a single oral dose of AZD5004 under fasted conditions.
  Interventions: Drug: AZD5004
- Group 2 (Experimental): Participants with normal renal function will receive a single oral dose of AZD5004 under fasted conditions.
  Interventions: Drug: AZD5004
- Group 3 (Optional) (Experimental): Participants with moderate renal impairment will receive a single oral dose of AZD5004 under fasted conditions.
  Interventions: Drug: AZD5004

INTERVENTIONS:
Drug: AZD5004 — Dose 1
  Other Names: ECC5004; Dose 1

SUMMARY:
This is a Phase I, multicentre, single-dose, non-randomised, open-label, parallel-group study to examine the PK, safety, and tolerability of AZD5004 in male and female participants with severe renal impairment and moderate renal impairment (optional) compared with male and female participants with normal renal function.

DETAILED DESCRIPTION:
This is a Phase I, multicentre, single-dose, non-randomised, open-label, parallel-group study to examine the PK, safety, and tolerability of AZD5004 in male and female participants with severe renal impairment and moderate renal impairment (optional) compared with male and female participants with normal renal function.

Participants will be assigned to the following groups based on eGFR determined at screening by a local laboratory using serum creatinine:

Group 1: Participants with severe renal impairment (eGFR < 30 mL/min), not on dialysis.

Group 2: Participants with normal renal function (eGFR of ≥ 90 mL/min) matched by sex, age, and body weight on a group level to the impaired participants.

Group 3 (optional): Participants with moderate renal impairment (eGFR ≥ 30 to < 60 mL/min).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-80 years of age
* Weight >50kg and BMI between 18-40 kg/m2

For participants with normal renal function:

-Participant must be medically healthy with no significant findings on medical evaluation and an eGFR ≥90 ml/min at screening.

For participants with renal impairment:

Group 1 (severe) must have an eGFR <30 ml/min and Group 3 (moderate) must have an eGFR 30 to <60 ml/min based on CKD-EPI calculations for at least 6 months prior to enrollment.

Exclusion Criteria:

* Poorly controlled diabetes mellitus (A1C >10% at screening or recent history of diabetic ketoacidosis or symptomatic hypoglycemia).
* Unwillingness to use adequate contraception
* Uncontrolled hypertension or hypotension.
* Positive screening for HIV, Hepatitis B, or Hepatitis C
* Presence of unstable systemic disease or psychologic conditions. Abnormal laboratory values to include but not limited to liver function tests (thresholds differ for renal impairment and health controls)
* Any change in baseline medication within 2 weeks of planned study initiation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
AUCinf | Day 1 to Day 5
  Area under the concentration-time curve from zero to infinity
AUClast | Day 1 to Day 5
  Area under the concentration-time curve from zero to the last measurable concentration
Cmax | Day 1 to Day 5
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Tmax | Day 1 to Day 5
  Time to reach maximum observed plasma concentration
PK parameter t1/2λz | Day 1 to Day 5
  Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve
PK parameter CL/F | Day 1 to Day 5
  Apparent total body clearance of drug from plasma after extravascular administration
PK parameter CLNR/F | Day 1 to Day 5
  non-renal clearance of drug from plasma after oral administration
PK parameter Vz/F | Day 1 to Day 5
  Apparent volume of distribution during the terminal phase after extravascular administration
PK parameter CLr | Day 1 to Day 5
  Renal clearance of the drug from plasma
PK parameter Ae | Day 1 to Day 5
  Cumulative amount of unchanged drug excreted into the urine
fe | Day 1 to Day 5
  Fraction of the drug excreted into the urine

OTHER OUTCOMES:
Number of participants with adverse events (AEs) | Day 1 to Day 10
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with severe and moderate (optional) renal impairment and those with normal renal function
Number of participants with abnormal Vital signs, abnormal ECGs, and abnormal physical examination findings | Day 1 to Day 5
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with severe and moderate (optional) renal impairment and those with normal renal function
Number of participants with abnormal laboratory tests results | Day 1 to Day 5
  To assess the safety and tolerability of a single oral dose of AZD5004 for participants with severe and moderate (optional) renal impairment and those with normal renal function

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home